CLINICAL TRIAL: NCT00971997
Title: The Study of Stepwise Introduction of Insulin Analog Mixture as a Post-marketing Clinical Trial of Lispro Mix 50/50 to Evaluate Efficacy and Safety in Type 2 Diabetic Patients With Inadequate Glycemic Control on Oral Therapy. (SIMPLE Study)
Brief Title: A Study of Insulin Lispro Mix in Type 2 Diabetic Asian Patients
Acronym: SIMPLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13329; F3Z-JE-IOPU (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-09-02; First posted 2009-09-04 (Estimated); Results first posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — isophane insulin, insulin lispro drug combination 50:50; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lispro 50/50 (Experimental)
  Interventions: Drug: Lispro Mix 50/50

INTERVENTIONS:
Drug: Lispro Mix 50/50 — Administered subcutaneously once daily for 16 weeks, twice daily for 16 weeks, and three times daily for 16 weeks dependent on glycemic control.
  Other Names: LY275585; Humalog Mix50

SUMMARY:
The purpose is to evaluate the proportion of subjects achieving a Hemoglobin A1c (HbA1c) level below 6.5%, when lispro mix 50/50 is introduced in a stepwise manner from every day (QD) administration to type 2 diabetic patients who have failed to achieve adequate glycemic control on oral antidiabetic drugs (OADs).

DETAILED DESCRIPTION:
A multicenter, non-randomized, open-label, post-marketing clinical study. The target population of the study is type 2 diabetic patients who have failed to achieve adequate glycemic control on OADs. The study consists of 4 periods: Lead-in Period (2 to 4 weeks), Study Period I (16 weeks), Study Period II (16 weeks), and Study Period III (16 weeks). The regimen of lispro mix 50/50 injection will be changed every 16 weeks based on the HbA1c level. During Study Period I, all the subjects will be given a once daily (QD) injection of lispro mix 50/50. During Study Period II, the regimen of lispro mix 50/50 injection will be changed to twice daily (BID) if the HbA1c level at Week 16 is 6.5% or above, and QD injection will be continued if the value is below 6.5%. During Study Period III, if the HbA1c level at Week 32 is 6.5% or above, the subjects on BID treatment during the previous period (Study Period II) will receive three times daily (TID) injections of insulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having type 2 Diabetes.
* Patients who have not been on insulin treatment within 6 months.
* Patients who have been taking OADs for at least 90 days.
* Patients with an HbA1c level in the range of 7.5% to 11.0%.
* Patients with a Body-Mass Index (BMI) of 35 kg/m² or below.

Exclusion Criteria:

* Patients having pre-proliferative or proliferative retinopathy (except for old retinopathy with no need for treatment).
* Patients having or suspected of having malignancy
* Patients having serious complications of the heart, liver, or kidney.
* Patients hypersensitive or allergic to insulin or insulin analog preparations or a history of it.
* Patients receiving systemic steroids.
* Are currently enrolled in a clinical trial of a non-approved drug. Or patients who participated in other clinical trials including post-marketing clinical trials within 90 days prior to informed consent being obtained.
* Patients of child-bearing potential. Breastfeeding patients. Patients with a positive result in a pregnancy test performed for women of child-bearing potential.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Japan (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamanashi

RESULTS

PARTICIPANT FLOW:
Groups:
- Lispro 50/50: Administered subcutaneously once daily for 16 weeks, twice daily for 16 weeks, and three times daily for 16 weeks dependent on glycemic control
Period: Overall Study
Arm/Group | Lispro 50/50
Started | 135
Completed | 116
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
Age Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 135
Region of Enrollment [Number; unit: participants]
  Japan | 135

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hemoglobin A1c (HbA1c) Below 6.5% at Week 48 Endpoint
Description: Hemoglobin A1c (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The 6.5% HbA1c is the Japan Diabetes Society (JDS) value, and is equivalent to the National Glycohemoglobin Standardization Program (NGSP) HbA1c value of 6.9%.
Time Frame: Week 48
Population: Participants received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
percentage of participants | 18.5 [12.4 to 26.1]

2. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c (HbA1c) Below 6.5% at Week 16 and Week 32 Endpoints
Description: as for outcome 1
Time Frame: Week 16 and Week 32
Population: Participants received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
percentage of participants
  Week 16 | 6.7 [3.1 to 12.3]
  Week 32 | 20.0 [13.6 to 27.7]

3. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c (HbA1c) Below 7.0% at Week 16, 32 and 48 Endpoints
Description: Hemoglobin A1c (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. The 7.0% HbA1c is the Japan Diabetes Society (JDS) value, and is equivalent to the National Glycohemoglobin Standardization Program (NGSP) HbA1c value of 7.4%.
Time Frame: Week 16 and Week 32 and Week 48
Population: Participants received at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
percentage of participants
  Week 16 | 22.2 [15.5 to 30.2]
  Week 32 | 43.0 [34.5 to 51.8]
  Week 48 | 52.6 [43.8 to 61.2]

4. Secondary Outcome: Percentage of Participants Achieving Hemoglobin A1c (HbA1c) Level Below 6.5% and Below 7.0% by Regimen at Week 48 Endpoint
Description: Hemoglobin A1c (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. 6.5% and 7.0% HbA1c are the Japan Diabetes Society (JDS) values, and are equivalent to the National Glycohemoglobin Standardization Program (NGSP) HbA1c values of 6.9% and 7.4%, respectively.
Time Frame: Week 48
Population: Participants completed treatment through Week 48.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Lispro 50/50 Once Daily; Lispro 50/50 Twice Daily; Lispro 50/50 Three Times Daily: Administered subcutaneously once daily for 16 weeks, twice daily for 16 weeks, and three times daily for 16 weeks dependent on glycemic control
Arm/Group | Lispro 50/50 Once Daily | Lispro 50/50 Twice Daily | Lispro 50/50 Three Times Daily
Number analyzed (Participants) | 9 | 21 | 86
percentage of participants
  Below 6.5% | 22.2 [2.8 to 60] | 61.9 [38.4 to 81.9] | 11.6 [5.7 to 20.3]
  Below 7.0% | 77.8 [40.0 to 97.2] | 95.2 [76.2 to 99.9] | 51.2 [40.1 to 62.1]

5. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 48 Endpoint
Description: Hemoglobin A1c (HbA1c) is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, Week 48
Population: Participants received at least one dose of the study drug, and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 134
percentage of glycosylated hemoglobin | -1.27 (0.98)

6. Secondary Outcome: Change From Baseline in Fasting Glucose at Week 48 Endpoint
Time Frame: Baseline, Week 48
Population: Participants received at least one dose of the study drug, and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 131
milligram/deciliter (mg/dL) | -19.9 (48.3)

7. Secondary Outcome: Change From Baseline in Blood Glucose Profile at Week 48 Endpoint
Description: Time course of changes in blood glucose was determined by 7-point self-monitoring of blood glucose (SMBG) during the day (before breakfast, lunch, and dinner, 2 hours after the start of each meal, and at bedtime).
Time Frame: Baseline, Week 48
Population: Participants received at least one dose of the study drug, and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 116
mg/dL
  Before breakfast (n=100) | -25.4 (55.0)
  After breakfast (n=98) | -58.6 (87.6)
  Before lunch (n=100) | -40.6 (73.1)
  After lunch (n=99) | -44.0 (84.5)
  Before dinner (n=100) | -40.0 (76.8)
  After dinner (n=97) | -55.9 (96.7)
  Bedtime (n=91) | -56.6 (75.3)

8. Secondary Outcome: Change From Baseline in Fasting C-Peptide at Week 48 to Endpoint
Description: C-peptide is a protein that is produced in the body along with insulin.
Time Frame: Baseline, Week 48
Population: Participants received at least one dose of the study drug, and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 131
nanogram/milliliter (ng/mL) | -0.339 (0.739)

9. Secondary Outcome: Change From Baseline in Fasting Serum Lipids at Week 48 Endpoint
Time Frame: Baseline, Week 48
Population: Participants received at least one dose of the study drug, and had both baseline and post-baseline values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
mg/dL
  Total cholesterol (n=131) | 1.6 (25.2)
  High-density lipoprotein (HDL) cholesterol (n=130) | 2.44 (8.66)
  Triglycerides (n=131) | -0.5 (70.4)

10. Secondary Outcome: Change From Baseline in Body Weight at Week 48 Endpoint
Time Frame: Baseline, Week 48
Population: Participants who completed treatment through Week 48, and had both baseline and post-baseline value.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 116
kilogram (kg) | 1.51 (3.18)

11. Secondary Outcome: Total Daily Dose of Insulin at Baseline, Week 16, Week 32 and Week 48
Time Frame: Baseline and Weeks 16, 32 and 48
Population: Participants who completed treatment through Week 48.
Measure: Mean (Standard Deviation); unit: units of insulin/day
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 116
units of insulin/day
  Baseline | 4.34 (1.35)
  Week 16 | 9.94 (4.91)
  Week 32 | 15.92 (10.01)
  Week 48 | 19.42 (13.64)

12. Secondary Outcome: Percentage of Participants Developing Hypoglycemia at Any Time From Baseline Through Week 48
Description: Results are reported as the percentage of participants experiencing hypoglycemia, which was considered any hypoglycemic event in which participants themselves recognized hypoglycemia-related signs and symptoms, or they had a blood glucose level below 50 milligram/deciliter (mg/dL) regardless of signs, symptoms or the relationship to treatment.
Time Frame: Baseline through Week 48
Population: Participants received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
percentage of participants | 65.9

13. Secondary Outcome: Number of Hypoglycemia Episodes Participants Experienced at Any Time From Baseline Through Week 48
Description: A hypoglycemic episode was considered any hypoglycemic event in which participants themselves recognized hypoglycemia-related signs and symptoms, or participants had a blood glucose level below 50 mg/dL regardless of signs, symptoms or the relationship to treatment.
Time Frame: Baseline through Week 48
Population: Participants received at least one dose of the study drug.
Measure: Number; unit: number of hypoglycemic episodes
Arm/Group | Lispro 50/50
Number analyzed (Participants) | 135
number of hypoglycemic episodes | 535

ADVERSE EVENTS:
Arm/Group | Lispro 50/50
Serious Adverse Events (participants affected / at risk) | 7/135
Other Adverse Events (participants affected / at risk) | 106/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lispro 50/50 (N=135)
Angina pectoris (Cardiac disorders) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lispro 50/50 (N=135)
Diabetic retinopathy (Eye disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 8 (9)
Seasonal allergy (Immune system disorders) | 6 (6)
Gastroenteritis (Infections and infestations) | 5 (6)
Nasopharyngitis (Infections and infestations) | 44 (58)
Contusion (Injury, poisoning and procedural complications) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 5 (7)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days